CLINICAL TRIAL: NCT04536298
Title: A Cluster-Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy of Vitamin D3 Supplementation to Reduce Disease Severity in Persons With Newly Diagnosed COVID-19 Infection and to Prevent Infection in Household Members
Brief Title: Vitamin D for COVID-19 Trial
Acronym: VIVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Harvard School of Public Health (HSPH) (Other); Fenway Health and Beth Israel Deaconess Medical Center (Unknown); Tishcon Corporation (Unknown); Takeda (Industry); Quest Diagnostics-Nichols Insitute (Industry); Laboratory Corporation of America (Industry); Trialfacts (Unknown); Karolinska Institutet (Other); Philanthropic donations (Unknown)
Responsible Party: Principal Investigator, JoAnn E. Manson, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002815
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2 infection; coronavirus; vitamin D; hospitalization; death; disease severity; treatment; prevention
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Death | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D (Active Comparator): Daily vitamin D3 (9600 IU/day on days 1 and 2; 3200 IU/day on days 3 through 28)
  Interventions: Dietary Supplement: vitamin D
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D — Vitamin D softgel capsules; each capsule contains 3200 IU of vitamin D3. Three capsules per day (9600 IU/day) will be taken on days 1 and 2, and one capsule per day (3200 IU/day) will be taken on days 3 through 28
  Other Names: vitamin D3; cholecalciferol
  Arms: Vitamin D
Dietary Supplement: Placebo — Placebo softgel capsules. Three capsules per day will be taken on days 1 and 2, and one capsule per day will be taken on days 3 through 28
  Arms: Placebo

SUMMARY:
The Vitamin D for COVID-19 Trial (VIVID) is a randomized, placebo-controlled clinical trial in 2024 men and women from across the U.S. and Mongolia to investigate whether taking a daily dietary supplement of vitamin D vs. placebo for 4 weeks reduces the rate of seeking healthcare for symptoms or concerns related to COVID-19 in participants recently diagnosed with COVID-19, and reduces the risk of infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in household contacts of individuals with newly diagnosed COVID-19.

DETAILED DESCRIPTION:
Data from laboratory studies, epidemiologic research, and randomized clinical trials conducted in the pre-COVID era strongly suggest that vitamin D is active in pathways relevant to immune function and may reduce the risk of acute respiratory infections. More recently, some observational studies have shown a significant association between low vitamin D status and worse clinical outcomes among COVID-19 patients. Whether vitamin D supplementation can reduce the risk of adverse clinical outcomes in recently diagnosed COVID-19 patients and/or reduce risk of infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV- 2) in those likely to have been exposed to the virus (post-exposure prophylaxis) is unknown.

The Vitamin D for COVID-19 Trial (VIVID) is a pragmatic, cluster-randomized clinical trial in 2024 men and women recruited nationwide from the U.S. and Mongolia. The trial is investigating whether taking a daily dietary supplement of vitamin D3 vs. placebo for 4 weeks reduces the rate of seeking healthcare visits (including hospitalizations, emergency room visits, or ambulatory or virtual clinician visits) for symptoms or concerns related to COVID-19 or deaths in people newly diagnosed with COVID-19, and reduces the risk of SARS-CoV-2 infection in household contacts of individuals with newly diagnosed COVID-19.

The trial has enrolled 1747 individuals aged 18 or older who are newly diagnosed with COVID-19 ("index cases") and 277 household contacts aged 18 or older.

Following receipt of informed consent, participants are randomized -- i.e., assigned by chance (like a coin toss) -- to one of two groups: (1) daily vitamin D3 (9600 IU/day on days 1-2; 3200 IU/day on days 3-28) or (2) daily vitamin D placebo. Index cases and household contacts of an index case (limited to at most one contact per household), if any, are assigned to the same group (cluster randomization). Participants take three oral softgel capsules on day 1, three capsules on day 2, and one capsule each day on days 3 through 28. Participants receive a 4-week supply of study capsules via overnight courier service.

Participants fill out a short (15-20 minute) questionnaire each week during the 4-week pill-taking period, as well as a follow-up questionnaire at 8 weeks after randomization. These questionnaires ask about symptoms, general health, and use of medications and dietary supplements. Questionnaires are completed online using a secure Internet-based system known as the Research Electronic Data Capture (REDCap) system. Participants must have an e-mail address to enroll in the study. Occasionally, participants (or their delegates) may receive a telephone call from study staff to collect information or to clarify answers on the questionnaire. Participants may contact investigators or staff using a toll-free number, if they have any questions or need assistance.

Participants (or their delegates) who indicate on a study questionnaire that they have been hospitalized are sent a medical release form to be signed and returned. The release form is used to get medical records from the participant's physician or hospital to confirm the specific reason for the hospitalization. In the event of a participant's death, the participant's delegate is sent a medical release form to be signed and returned. The release form is used to get medical records from the participant's physician or hospital to confirm the specific cause of death.

Participants provide dried blood spot samples at baseline and week 4. Participants provide these samples using a sample collection kit mailed to their homes. Blood samples are collected through a finger prick onto a filter paper. Blood samples are stored and will be used to measure vitamin D (25(OH)D) levels. A subsample of participants provide follow-up dried blood spot samples at weeks 1, 2, or 3 to clarify the time course of 25(OH)D increase. In participants who are not diagnosed with COVID-19 during the study, blood samples will also be tested for COVID-19 antibodies.

Support for VIVID is provided by Harvard University and private philanthropy. Tishcon Corporation (Salisbury, Maryland, USA) is donating the study capsules. The Karolinska Institute (Stockholm, Sweden) is donating the serology assessment.

ELIGIBILITY:
Inclusion/exclusion criteria for INDEX CASES:

Inclusion criteria

1. Adults aged 18 years or older who are newly diagnosed with COVID-19 infection within 7 days of testing.
2. Ability and willingness to understand and provide informed consent.

Exclusion criteria

1. Known current pregnancy.
2. Current hospitalization.
3. Unable to complete online questionnaires or adhere to study requirements.
4. Consume more than 1000 IU per day of vitamin D from all supplemental sources combined (individual vitamin D supplements, calcium plus vitamin D supplements, medications with vitamin D [e.g., Fosamax Plus D], and multivitamins) in the past 4 weeks.
5. Use of prescription vitamin D treatments (Calcitriol [Rocaltrol, Calcitrol, Vectical, Calcijex] or Paricalcitol [Zemplar]).
6. Consume supplements with more than 1200 mg calcium per day.
7. Known diagnosis of hypercalcemia or a condition associated with vitamin D hypersensitivity.
8. Prior diagnosis of cancer *AND* currently undergoing radiation, chemotherapy, or immunotherapy.
9. Kidney failure or dialysis; severe liver disease or cirrhosis.
10. Any parathyroid conditions.
11. Use of medications for seizures or epilepsy. Examples: Carbamazepine (Carbatrol, Tegretol), Phenytoin (Dilantin, Phenytek), Valproic acid (Depakene), Oxcarbazepine (Oxtellar, Trileptal), Phenobarbital, Topiramate (Topamax).
12. Use of digoxin.
13. Inability to receive an overnight express mail shipment of study pills at a home address.
14. Participation in other COVID-19 trials.

Inclusion/exclusion criteria for HOUSEHOLD CONTACTS:

Inclusion criteria:

1. Persons aged 18 years or older who live in the same household with an index individual and have been identified as the closest household contact within the same household (limited to 1 per household).
2. Persons aged 18 years or older who live in household with someone who tested positive for COVID-19 within past 7 days but not participating in VIVID.
3. Ability and willingness to understand and provide informed consent.

Exclusion criteria:

1. Known current pregnancy.
2. History of SARS-CoV-2 infection.
3. Receipt of a SARS-CoV-2 vaccination or monoclonal antibody.
4. Unable to complete online questionnaires or adhere to study requirements.
5. Consume more than 1000 IU per day of vitamin D from all supplemental sources combined (individual vitamin D supplements, calcium plus vitamin D supplements, medications with vitamin D [e.g., Fosamax Plus D], and multivitamins) in the past 4 weeks.
6. Use of prescription vitamin D treatments (Calcitriol [Rocaltrol, Calcitrol, Vectical, Calcijex] or Paricalcitol [Zemplar]).
7. Consume supplements with more than 1200 mg calcium per day.
8. Known diagnosis of hypercalcemia or a condition associated with vitamin D hypersensitivity.
9. Prior diagnosis of cancer *AND* currently undergoing radiation, chemotherapy, or immunotherapy.
10. Kidney failure or dialysis; severe liver disease or cirrhosis.
11. Any parathyroid condition.
12. Use of medications for seizures or epilepsy. Examples: Carbamazepine (Carbatrol, Tegretol), Phenytoin (Dilantin, Phenytek), Valproic acid (Depakene), Oxcarbazepine (Oxtellar, Trileptal), Phenobarbital, Topiramate (Topamax).
13. Use of digoxin.
14. Inability to receive an overnight express mail shipment of study pills at a home address.
15. Participation in other COVID-19 trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2024 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of seeking healthcare visits (including hospitalizations, emergency room visits, or ambulatory or virtual clinician visits) for symptoms or concerns related to COVID-19 or deaths in participants newly diagnosed with COVID-19 (index cases) | 4 weeks

SECONDARY OUTCOMES:
Rate of in-person healthcare visits related to COVID-19 infection among index cases | 4 weeks
Disease symptom score in index cases | 4 weeks
  Area under curve (AUC) of weekly self-reported symptom score (summed across all symptoms) through week 4
Disease severity in index cases | 4 weeks
  Self-report of at least one severe symptom
Time to seeking healthcare (including hospitalizations, emergency room visits, or ambulatory or other clinician visits) or death in index cases | 4 weeks
SARS-CoV-2 infection in close household contacts | 4 weeks
  Self-report of positive test
Long COVID symptoms in index cases | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn E Manson, MD, DrPH, Principal Investigator — Brigham and Women's Hospital; Rui Wang, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM); Davaasambuu Ganmaa, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Details will be provided at a later date.

REFERENCES:
- [Background] Manson JE, Bassuk SS. Commentary. Eliminating vitamin D deficiency during the COVID-19 pandemic: A call to action. Metabolism. 2020 Nov;112:154322. doi: 10.1016/j.metabol.2020.154322. Epub 2020 Jul 23. No abstract available. PMID 32712223
- [Background] Wang R, DeGruttola V, Lei Q, Mayer KH, Redline S, Hazra A, Mora S, Willett WC, Ganmaa D, Manson JE. The vitamin D for COVID-19 (VIVID) trial: A pragmatic cluster-randomized design. Contemp Clin Trials. 2021 Jan;100:106176. doi: 10.1016/j.cct.2020.106176. Epub 2020 Oct 10. PMID 33045402